CLINICAL TRIAL: NCT01015209
Title: Safety and Tolerability of Chitosan-N-acetylcysteine Eye Drops in Healthy Young Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT- 141009
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: 18 healthy subjects (Active Comparator): 18 healthy subjects receiving Chitosan- N- Acetylcysteine eye drops at a dose of 0.1%, 0.2% or 0.3% (6 subjects per group)
  Interventions: Device: Chitosan- N- Acetylcysteine eye drops
- Cohort 2: 12 healthy patients (Active Comparator): 12 healthy subjects receiving Chitosan- N- Acetylcysteine eye drops at a dose of 0.1%, 0.2% or 0.3%
  Interventions: Device: Chitosan- N- Acetylcysteine eye drops

INTERVENTIONS:
Device: Chitosan- N- Acetylcysteine eye drops — Cohort 1: 1 drop once Cohort 2: 2 drops daily for 5 days

SUMMARY:
The "dry eye syndrome" DES is a highly prevalent ocular disease, in particular in the elderly population. One mainstay of therapy for patients suffering from DES is the use of topically administered lubricants. However, despite many efforts, no "ideal" formulation has yet been found.

Recently, Croma Pharma has introduced chitosan-N-acetylcysteine eye drops, designed for treatment of symptoms related to DES. Chemically, chitosan is a polycationic biopolymer with favourable biological properties such as high biocompatibility and low toxicity. Additionally, the new formulation comprises N-acetylcysteine, which has been used in ophthalmology because of its mucolytic properties for several years. Based on theoretical considerations, one can hypothesize that the new chitosan derivative may show an increased adhesion to mucins of the ocular surface and may therefore be particularly beneficial in reducing the symptoms associated with DES.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 45 years
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 dpt.

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Abuse of alcoholic beverages
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ametropia of 6 or more dpt.
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Difference between the treated and the non- treated eye with Chitosan- N- Acetylcysteine eye drops | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria